CLINICAL TRIAL: NCT01052051
Title: Clinical Trial of Vitamin D3 to Reduce Cancer Risk in Postmenopausal Women
Acronym: CAPS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joan Lappe, Professor of Nursing and Medicine, Creighton University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAPS08-15024; R01CA129488-01A2 (NIH)
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D3 and calcium carbonate (Experimental): Daily vitamin D3 2000 IU/day and calcium carbonate 1500mg/day supplementation
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate
- Placebo for vitamin D3 and calcium carbonate (Placebo Comparator): Placebo for daily vitamin D3 and calcium carbonate
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 2000 IU/daily
Dietary Supplement: Calcium carbonate — Calcium carbonate 1500mg / daily

SUMMARY:
To determine the effect of increasing serum 25(OH)D from prevailing levels with vitamin D3 supplementation, while maintaining adequate calcium intake, on incidence of all-type cancer in a population sample of healthy postmenopausal women.

DETAILED DESCRIPTION:
Hypotheses:

Primary: Increasing serum 25(OH)D from prevailing levels with vitamin D3 supplementation, while maintaining adequate calcium intake, will significantly decrease incidence of all-type cancer in a population sample of healthy postmenopausal women.

Secondary:

1. Increasing serum 25(OH)D from prevailing levels will significantly decrease incidence of specific cancers: breast, lung, colon, myeloma, leukemia, lymphoma.
2. Increasing serum 25OHD from prevailing levels will significantly decrease incidence of other disorders, specifically hypertension, cardiovascular disease, osteoarthritis, colonic adenomas, diabetes, upper respiratory infections and falls.

Specific Aims:

1. Determine the effect of supplementation with vitamin D3 on incidence of all types of cancer combined.
2. Determine in a nested-case control study the association of serum 25OHD collected at randomization and at the end of year one of study with risk of cancer over four years.
3. Sample randomly the population of healthy independently-living postmenopausal women 55 years and older from twelve adjacent rural counties in Nebraska.
4. Enroll a random sample of 2300 women into an intervention study, assign them randomly to one of two treatment groups: 1) vitamin D3 (2000 IU/d) and calcium (1500 mg/d), or 2) vitamin D3 placebo and calcium placebo, and to follow each study participant for four years.
5. Collect and store blood serum and white blood cells from every participant to test for genetic markers should the intervention be found effective in decreasing the incidence of cancer. Markers selected will be determined by the state of the science at the time of analysis.
6. Determine the effect of supplementation with calcium and vitamin D3 on incidence of specific cancers: breast, lung, colon, myeloma, leukemia, and lymphoma.
7. Determine the effect of supplementation on incidence of other disorders, specifically hypertension, cardiovascular disease, osteoarthritis, colonic adenomas, diabetes, upper respiratory infections, fractures, and falls.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 55 years
* Last menstrual period (LMP): ≥ 4 years
* Good general health
* Willingness to participate in this 4 year long study
* Able to give informed consent
* Able to live independently and travel to the Fremont Area Medical Center (FAMC) for study visits

Exclusion Criteria:

* History of cancer except

  * Superficial basal or squamous cell carcinoma of the skin
  * Other malignancies treated curatively more than 10 years ago
* History of renal calculi or chronic kidney disease
* History of sarcoidosis
* History of tuberculosis
* Participation in the previous Creighton cancer prevention study
* Mini-Mental Status Exam (MMSE) score of ≤ 23. Use the MMSE if there are any concerns about the person's cognitive abilities or ability to give fully informed consent to the study. Concerns may be related to a person's lack of orientation to person, place, or time; language difficulties (inability to structure simple, complete sentences); or short term memory. The Hartford Institute for Geriatric Nursing recommends that a score of 23 or lower indicates cognitive impairment. (Accessed at www.harforddign.org). See appendix.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2303 (Actual)
Dates: Start 2009-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
all-type cancer (excluding non-melanoma skin cancers) | 4 years

SECONDARY OUTCOMES:
breast cancer | 4 years
colorectal cancer | 4 years
new osteoporotic fractures | 4 years
diagnosis of diabetes mellitus | 4 years
frequency and severity of asthma symptoms in persons with asthma at baseline | 4 years
frequency of falls | 4 years
frequency of colds and flu | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Joan M Lappe, PhD, Principal Investigator — Creighton University
Locations (1):
- Fremont Area Medical Center, Fremont, Nebraska, United States

REFERENCES:
- [Derived] Lappe J, Watson P, Travers-Gustafson D, Recker R, Garland C, Gorham E, Baggerly K, McDonnell SL. Effect of Vitamin D and Calcium Supplementation on Cancer Incidence in Older Women: A Randomized Clinical Trial. JAMA. 2017 Mar 28;317(12):1234-1243. doi: 10.1001/jama.2017.2115. PMID 28350929